CLINICAL TRIAL: NCT00807261
Title: PhaseⅡ Study of Weekly Docetaxel and Fixed-Dose Rate Gemcitabine in Patient With Previously Treated Advanced Soft Tissue and Bone Sarcoma Prospective, Open Label, Multi-Institutional
Brief Title: Weekly Docetaxel and Fixed-Dose Rate Gemcitabine Combination Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Asan Medical Center (Other)
Collaborators: Severance Hospital (Other); Korea University Anam Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Jin-hee Ahn / Associate Professor, AMC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DOCET_L_03981
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine and Docetaxel — Drug and schedule
  * Gemcitabine 1000 mg/m2 IV over 10 mg/m2/min (D1, D8)
  * Docetaxel 35 mg/m2 IV (D1, D8) .. every 21 days
  Dose modification
  * Treatment should be delayed if the ANC<1,500/ mm3, or if the platelet count <75,000/mm3 on the first day of the next cycle.
  * Gemcitabine & docetaxel are omitted on day 8, when ANC is less than 1000/mm3 or platelet count is less than 50,000/mm3; it is reduced by 25% if the ANC is between 1,000 and 1,500/mm3 or the platelet count is between 50,000 and 75,000/mm3 Study design Treatment should consist of at least 2 cycles unless rapid disease progression or unacceptable toxicities occur after one cycle of chemotherapy.
  Patients with response or no change will receive 2 additional cycles.

SUMMARY:
To determine the activity of weekly Docetaxel and Gemcitabine in patients with advanced soft tissue sarcoma previously treated with anthracycline and/or ifosfamide

1. Primary endpoint: response rate
2. Secondary endpoint: progress-free survival, overall survival, safety

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic, unresectable soft tissue sarcoma or bone sarcoma with the exception of certain histopathologic subtypes of sarcomas recognized by experts to derive no benefit from conventional chemotherapy (e.g., alveolar soft part sarcoma, clear cell sarcoma, chondrosarcoma, chordoma, desmoid tumors)
* Bone sarcoma patients must have visceral metastatic disease (e.g., metastatic to lung or liver)
* Patients who were previously treated with anthracycline- and/or ifosfamide- containing chemotherapy, as a first-line chemotherapy for metastatic disease, or adjuvant therapy Patients may have had up to 2 prior chemotherapies within 4 weeks of starting the study treatment
* unidimensional measurable lesions
* Age ≥ 16 years
* Life expectancy of more than 3 months
* ECOG performance status ≤ 2
* Adequate bone marrow function (ANC≥1,500/mm3, and platelet count ≥100,000/mm3)
* Adequate kidney function (serum creatinine ≤ 1.5 mg/dL)
* Adequate liver function (bilirubin ≤ 2 mg/dl and transaminase level ≤ 3 times the upper normal limit, or < 5 times for patients with liver metastasis, serum alkaline phosphatase < 2.5 times the upper normal limit, or < 5 times if liver metastases were present or < 10 times if bone metastases were present).
* Adequate cardiac function (Ejection fraction ≥ 50% by echoCG or MUGA scan)
* All patients are fully informed about the nature and purpose of this study and should give informed consent before the start of treatment.

Exclusion Criteria:

* Pregnant or lactating patients
* Patients with resectable lung metastasis
* Presence or history of CNS metastasis
* Prior history of other cancer within past 5 years, asides from basal cell and squamous cell carcinoma of skin, and carcinoma in situ of uterine cervix
* Any preexisting medical condition of sufficient severity to prevent full compliance with the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-hee Ahn, Principal Investigator — AIDS Malignancy Consortium